CLINICAL TRIAL: NCT05562349
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2a Pilot Study to Assess the Efficacy and Safety of Clavulanic Acid vs. Placebo for the Treatment of Cocaine Use Disorder
Brief Title: Clavulanic Acid for the Treatment of Cocaine Use Disorder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: University of Pennsylvania (Other); Medical University of South Carolina (Other); Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 30076
Record Dates: First submitted 2022-09-15; First posted 2022-09-30 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Clavulanic Acid; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clavulanic Acid (Experimental): Participants may receive 500 mg of CLAV at baseline. Subjects who are using cocaine once per week or more and who can tolerate 500 mg/day for 4 weeks, will have a dose escalation to 750 mg/day. If tolerated, 750mg/day will be maintained for 8 weeks, otherwise the dose will decrease to 500mg/day.
  Interventions: Drug: Clavulanic Acid Only Product
- Placebo (Placebo Comparator): Participants may receive placebo and serve as a control group. They will be blinded to their condition and will have a "dose" escalation at the same time as the experimental group, and be given additional placebo pills to match the number given to the experimental group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clavulanic Acid Only Product — Drug will be given in 250mg capsules
  Other Names: Potassium clavulanate
  Arms: Clavulanic Acid
Drug: Placebo — Capsule with no active medication - identical to drug capsule
  Other Names: microcrystalline cellulose
  Arms: Placebo

SUMMARY:
A dose escalation study to assess the efficacy and safety of Clavulanic Acid (CLAV) vs. placebo (PBO) for the treatment of cocaine use disorder (CUD)

DETAILED DESCRIPTION:
This pilot study is indicated for treatment of moderate to severe cocaine use disorder. It is a randomized, placebo-controlled, parallel group, multi-center pilot study to compare the efficacy of 500-750mg/day clavulanic acid vs. placebo in addition to weekly medication management therapy. Subjective, cognitive, and adverse effect assessments, blood pressure and pulse will be performed 1-3 times weekly.

ELIGIBILITY:
Inclusion Criteria:

* Be able to verbalize understanding of consent form, able to provide written informed consent, and verbalize willingness to complete study procedures
* Be male or female adult volunteers ages 18-70 inclusive.
* Have a Diagnostic and Statistical Manual (DSM-V) diagnosis of cocaine use disorder, moderate to severe in early remission with a duration of regular (weekly or more) cocaine (either snorted, smoked or injected) for at least one year.
* Have a history and brief physical examination that demonstrate no clinically significant contraindication for participating in the study, and/ or significant or unstable medical or psychiatric illness.

Exclusion Criteria:

* Meets DSM-V criteria for dependence on any substance other than cocaine and mild to moderate alcohol or marijuana (except nicotine or caffeine), determined by the structured clinical interview for DSM-V.
* Allergy to clavulanic acid, penicillin, or any beta-lactam drug.
* Meets current or lifetime DSM-V criteria for schizophrenia or any psychotic disorder or organic mental disorder. Subject meets current DSM-V diagnosis of any other clinically significant psychiatric disorder that will interfere with study participation.
* Severe physical or medical illnesses such as AIDS or active hepatitis.
* If female, tests positive on a pregnancy test, is contemplating pregnancy in the next 6 months, is nursing, or is not using an effective contraceptive method (if relevant)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Changes in relapse to cocaine use in CLAV group vs PBO group | Last 3 weeks of 12 week study
  Cocaine-free weeks are measured by self-report using Timeline Follow Back (TLFB) and confirmed by urine drug screen.

SECONDARY OUTCOMES:
Changes in weekly abstinence in the CLAV group vs. PBO group | Self reported cocaine use and Urine Drug Screen (UDS) will be administered 1-3 times per week and at follow-up
  Abstinence from cocaine by week will be measured by self report and urine drug screen
Changes in weekly cocaine use will be greater in the CLAV group vs. PBO group | TLFB and UDS will be administered 1-3 times per week and at follow-up
  Cocaine-free visits are measured by self-report using TLFB confirmed by urine drug screen
Changes in subject health and function, quality-of-life, will be greater in the CLAV group vs. PBO group | Baseline, week 4, week 8, week 12
  Medical Outcomes Study Quality of Life Scale short form 36, will determine whether CLAV treatment is associated with improved QOL
Clavulanic acid 500-750 mg/day for 12 weeks will be safe and reasonably well tolerated | 1-3 times per week and at follow-up
  Safety and tolerability as assessed by the rates of occurrence of adverse events (AEs) and the severity
Cocaine craving will be decreased more by CLAV vs. PBO | 1-3 times per week and at follow-up
  Changes in craving will be greater in the CLAV group compared with PBO group, as measured by the cocaine craving questionnaire (CCQ), adjusted for baseline and sex

OTHER OUTCOMES:
Changes in withdrawal symptoms over weeks 1, 2, 3 will occur in CLAV vs PBO group | Weekly for 3 weeks
  Withdrawal symptoms will be measured using the Cocaine Selective Severity Assessment (CSSA)
Executive control will change more in the CLAV group compared with the PBO group after 12 weeks | Baseline, week 4, week 8, week 12
  Delay discounting will measure executive control
Adverse Childhood Experiences (ACE) may correlate with cocaine relapse | Baseline, week 12, follow-up
  Relationship between baseline scores from the ACE scale and abstinence outcomes in CLAV group will be compared to PBO group

CONTACTS AND LOCATIONS:
Overall Officials: Mary Morrison, MD, MS, Principal Investigator — Temple University
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MUSC, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim J, John J, Langford D, Walker E, Ward S, Rawls SM. Clavulanic acid enhances glutamate transporter subtype I (GLT-1) expression and decreases reinforcing efficacy of cocaine in mice. Amino Acids. 2016 Mar;48(3):689-696. doi: 10.1007/s00726-015-2117-8. Epub 2015 Nov 5. PMID 26543027